CLINICAL TRIAL: NCT01319084
Title: Development of a Versatile Intra-operative On-screen Audiovisual Mentoring System Using TileproTM Program for Robotic Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2010-0062
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ARMES group: Surgeons who watch Tilepro program before da Vinci Robotic Surgery.
- normal group: Surgeons who do not watch Tilepro program before da Vinci Robotic Surgery.

SUMMARY:
Considering the development of gastric cancer surgery using da Vinci Robotic Surgical System, the development of educational program needs to be achieved in Korea and this institute. Moreover, because of the large number of gastrectomy including robotic surgery for gastric cancer treatment, the investigators can provide high quality of educational program using da Vinci System. Therefore, the investigators wanted to create an innovative real-time training module, which can provide an intraoperative step-by-step guide to robotic surgical procedures. This technological project was named as Advanced Robotic Multi-display Educational System (ARMES).

DETAILED DESCRIPTION:
Considering the development of gastric cancer surgery using da Vinci Robotic Surgical System, the development of educational program needs to be achieved in Korea and this institute. Moreover, because of the large number of gastrectomy including robotic surgery for gastric cancer treatment, the investigators can provide high quality of educational program using da Vinci System. Therefore, the investigators wanted to create an innovative real-time training module, which can provide an intraoperative step-by-step guide to robotic surgical procedures. This technological project was named as Advanced Robotic Multi-display Educational System (ARMES).

The four-stages of ARMES development are as follows:

1. Standardization of the key steps of the selected procedure;
2. Preparation of well edited short video clips for each of the previously determined steps using our extensive library of videos of over 350 high quality robotic gastrectomies;
3. Production of a 3D animation of the key surgical steps;
4. Integration of the video segments into the da Vinci Robot system using TileproTM.

Through predetermined standardized segments of short operation video clips and 3D animation, the investigators are developing a versatile intra-operative on-screen audiovisual mentoring system using TileproTM program, which will improve surgeons' capabilities to perform complex robotic operations achieving quicker operation specific competency. It will help surgeons at initial state of robotic surgery in technical as well as oncological aspect for cancer surgery in detail and step-by-step. Finally this program can be applied to other robotic surgery and progressed to be a standard education program.

ELIGIBILITY:
Inclusion Criteria:

* Robotic surgery for primary early gastric cancer
* Distal gastrectomy with Billroth II anastomosis
* Age: 20~80 years old

Exclusion Criteria:

* Other malignancy and inflammatory diseases
* Disease associated with bleeding tendency
* Previous major abdominal surgery
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic in severance hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea